CLINICAL TRIAL: NCT04622449
Title: Assessment of Role of Iron Metabolism, Nutritional Deficiency, Gastrointestinal Loss, and Chronic Inflammation in the Etiopathogenesis of Anemia in Chronic Liver Disease
Brief Title: Etiopathogenesis of Anemia in Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IM/2020/1624
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Anemia; Chronic Liver Disease
Keywords: Gastro Intestinal Bleeding; Iron Deficiency Anemia; Cirrhosis; Anemia of Chronic disease; Nutritional deficiency
MeSH Terms: conditions — Anemia; Gastrointestinal Hemorrhage; Anemia, Iron-Deficiency; Fibrosis; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen Serum Samples to measure IL-1, IL-6, Hepcidin levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic liver disease with anemia: All patients with anemia as diagnosed by WHO criteria in patients with liver disease of any etiology.

SUMMARY:
Anemia is the most common complication of liver cirrhosis and is seen in 75% of cases. The etiology of anemia in liver disease is diverse and often multi-factorial. Given the diverse and sometimes multifactorial etiology of cirrhosis, it is difficult to determine the exact cause of anemia in these groups of patients. The most common type of anemia encountered in liver cirrhosis is normocytic normochromic anemia, attributable to the chronic inflammatory state. The key question in management of anemia in patients with liver disease which specific factor needs to be corrected to restore hemoglobin levels and improve overall clinical status and improve severity scores.

DETAILED DESCRIPTION:
Common causes of anemia include acute and chronic blood loss due to upper gastrointestinal (GI) bleeding, malnutrition, hemolysis, hypersplenism secondary to portal hypertension, and impaired coagulation. Alcohol causes anemia by its direct bone marrow toxicity, vitamin B12 and folate deficiency due to poor oral intake, and intestinal malabsorption. Treatment related anemia is seen in patients with chronic hepatitis C virus infection receiving ribavirin and interferon. Hepatitis associated aplastic anemia, characterized by pancytopenia and hypocellular bone marrow, is an entity seen concurrently with or within 6 months of infection with hepatotropic viruses such as hepatitis B, hepatitis C and Epstein-Barr virus. Acute and chronic blood loss from varices, portal hypertensive gastropathy and gastric antral vascular ectasia can give rise to iron-deficiency anemia, in which the picture is one of microcytic hypochromic anemia. Another common hematological abnormality seen in liver cirrhosis is macrocytosis. The causes of macrocytosis in liver cirrhosis are also multi factorial. Vitamin B12 and folate deficiency is also frequently seen in liver cirrhosis, particularly of alcoholic origin, due to malnutrition and increased intestinal permeability, and gut dysbiosis.

Patients with cirrhosis patients have a high incidence of sepsis which can trigger decompensation and may result in prolonged hospital stay and increased mortality. Many studies have estimated that about 30%-50% admissions of patients with cirrhosis have sepsis. Of those who don't have sepsis at presentation, about 15% patients admitted to hospital develop sepsis during the hospital stay. After infection develops, the patient may develop acute kidney injury (AKI), shock, encephalopathy or disseminated intravascular coagulation (DIC) further decreasing the chances of survival. Sepsis and the associated cytokines have a myelosuppressive effect and prevent the erythron from making blood cells. This results in an increase in ferritin as an inflammatory biomarker and alters iron metabolism by affecting the production of hepcidin in the liver. The worsening of anemia in patients with sepsis is well documented, and this is further impacted using drugs like antibiotics which trigger inflammation mediated suppression of the erythron and other hematopoietic precursors like megakaryocytes and leucoblasts.

In the study, after taking informed consent, participants will be evaluated for etiology of chronic liver disease with proper history, clinical examination and investigations which will include viral markers (HbsAg, Anti-HCV, Total anti-Hbc, AIH markers (Anti-nuclear antibody/ anti-smooth muscle antibody/anti- liver kidney microsomal antibody), serum ceruloplasmin, non-alcoholic fatty liver disease (NAFLD) work up and radiological investigations for cirrhosis. The severity of cirrhosis will be determined by Child-Pugh's and MELD/MELD-Na score.

To evaluate for anemia, following results would be noted: Complete hemogram with RBC indices, reticulocyte count and peripheral blood smear, RFT, LFT, INR, iron studies - serum iron, ferritin, total iron binding capacity and %transferrin saturation, serum vitamin B12, folate levels. Workup for hemolysis would include lactate dehydrogenase, serum haptoglobin, direct coombs test and plasma hemoglobin. Upper GI endoscopy findings will also be noted to evaluate the contribution of gastrointestinal blood loss in causing anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Either gender
3. Patients with chronic liver disease with anemia (Hemoglobin in Non-pregnant women (18 years of age and above) <12g/dl and in men <13g/dl

Exclusion Criteria:

1. Those who do not consent to participate in the study
2. Renal dysfunction (S. Creatinine ≥ 2mg/dL)
3. Pregnancy/Lactation
4. Post liver transplant patients
5. HIV infection
6. Patients who are on psychoactive drugs, like sedatives or antidepressants
7. Patients with uncontrolled sepsis
8. Patients who are too sick to carry out the protocol
9. Patients with ongoing active bleeding
10. Patients with known primary hematological disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic liver disease attending outpatient department of hepatology, admitted under hepatology department or emergency services
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Etiologies of anemia in patients with liver disease | 1 month
  Determine the prevalence of various etiologies of anemia in patients with liver disease
Correlation with liver disease severity | 1 month
  Association of liver disease severity as measured by MELD, MELD Na and CTP scores with severity of anemia

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Casas R, Jones EA, Moreno-Otero R. Spectrum of anemia associated with chronic liver disease. World J Gastroenterol. 2009 Oct 7;15(37):4653-8. doi: 10.3748/wjg.15.4653. PMID 19787828
- [Background] Premkumar M, Saxena P, Rangegowda D, Baweja S, Mirza R, Jain P, Bhatia P, Kumar G, Bihari C, Kalal C, Vyas T, Choudhury A, Sarin SK. Coagulation failure is associated with bleeding events and clinical outcome during systemic inflammatory response and sepsis in acute-on-chronic liver failure: An observational cohort study. Liver Int. 2019 Apr;39(4):694-704. doi: 10.1111/liv.14034. Epub 2019 Feb 7. PMID 30589495
- [Background] Nahon P, Nuraldeen R, Rufat P, Sutton A, Trautwein C, Strnad P. In alcoholic cirrhosis, low-serum hepcidin levels associate with poor long-term survival. Liver Int. 2016 Feb;36(2):185-8. doi: 10.1111/liv.13007. Epub 2015 Dec 6. PMID 26561367
- [Background] Mathurin SA, Aguero AP, Dascani NA, Prestera JA, Gianserra C, Londero E, Chiorra C. [Anemia in hospitalized patients with cirrhosis: prevalence, clinical relevance and predictive factors]. Acta Gastroenterol Latinoam. 2009 Jun;39(2):103-11. Spanish. PMID 19663083
- [Background] Stein J, Connor S, Virgin G, Ong DE, Pereyra L. Anemia and iron deficiency in gastrointestinal and liver conditions. World J Gastroenterol. 2016 Sep 21;22(35):7908-25. doi: 10.3748/wjg.v22.i35.7908. PMID 27672287
- [Background] Tan TC, Crawford DH, Franklin ME, Jaskowski LA, Macdonald GA, Jonsson JR, Watson MJ, Taylor PJ, Fletcher LM. The serum hepcidin:ferritin ratio is a potential biomarker for cirrhosis. Liver Int. 2012 Oct;32(9):1391-9. doi: 10.1111/j.1478-3231.2012.02828.x. Epub 2012 Jun 7. PMID 22676252
- [Background] Gkamprela E, Deutsch M, Pectasides D. Iron deficiency anemia in chronic liver disease: etiopathogenesis, diagnosis and treatment. Ann Gastroenterol. 2017;30(4):405-413. doi: 10.20524/aog.2017.0152. Epub 2017 May 3. PMID 28655976
- [Background] Alexopoulou A, Vasilieva L, Kanellopoulou T, Pouriki S, Soultati A, Dourakis SP. Presence of spur cells as a highly predictive factor of mortality in patients with cirrhosis. J Gastroenterol Hepatol. 2014 Apr;29(4):830-4. doi: 10.1111/jgh.12473. PMID 24325340
- [Background] Paternostro R, Kapzan L, Mandorfer M, Schwarzer R, Benedikt S, Viveiros A, Bauer D, Ferlitsch M, Zoller H, Trauner M, Ferlitsch A. Anemia and iron deficiency in compensated and decompensated cirrhosis: Prevalence and impact on clinical outcomes. J Gastroenterol Hepatol. 2020 Sep;35(9):1619-1627. doi: 10.1111/jgh.14988. Epub 2020 Feb 26. PMID 31972057
- [Background] Intragumtornchai T, Rojnukkarin P, Swasdikul D, Israsena S. The role of serum ferritin in the diagnosis of iron deficiency anaemia in patients with liver cirrhosis. J Intern Med. 1998 Mar;243(3):233-41. doi: 10.1046/j.1365-2796.1998.00290.x. PMID 9627161
- [Background] Vassiliadis T, Mpoumponaris A, Vakalopoulou S, Giouleme O, Gkissakis D, Grammatikos N, Soufleris K, Kakafika A, Tziomalos K, Patsiaoura K, Papanikolaou V, Evgenidis N. Spur cells and spur cell anemia in hospitalized patients with advanced liver disease: Incidence and correlation with disease severity and survival. Hepatol Res. 2010 Feb;40(2):161-70. doi: 10.1111/j.1872-034X.2009.00590.x. Epub 2010 Jan 11. PMID 20070401
- [Background] Liangpunsakul S, Ulmer BJ, Chalasani N. Predictors and implications of severe hypersplenism in patients with cirrhosis. Am J Med Sci. 2003 Sep;326(3):111-6. doi: 10.1097/00000441-200309000-00001. PMID 14501224
- [Background] Simbrunner B, Beer A, Woran K, Schmitz F, Primas C, Wewalka M, Pinter M, Dolak W, Scheiner B, Puespoek A, Trauner M, Oberhuber G, Mandorfer M, Reiberger T. Portal hypertensive gastropathy is associated with iron deficiency anemia. Wien Klin Wochenschr. 2020 Jan;132(1-2):1-11. doi: 10.1007/s00508-019-01593-w. Epub 2020 Jan 7. PMID 31912289
- [Background] Bothou C, Ruschenbaum S, Kubesch A, Quenstedt L, Schwarzkopf K, Welsch C, Zeuzem S, Welzel TM, Lange CM. Anemia and Systemic Inflammation Rather than Arterial Circulatory Dysfunction Predict Decompensation of Liver Cirrhosis. J Clin Med. 2020 Apr 26;9(5):1263. doi: 10.3390/jcm9051263. PMID 32357568